CLINICAL TRIAL: NCT04160039
Title: Early Cycle Ergometry for Critically-Ill Liver Failure Patients in a Transplant Intensive Care Unit
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left institution
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO32773
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Liver Cirrhoses; Liver Failure; ICU Acquired Weakness
Keywords: Cycle Ergometry; Physical Therapy; Rehabilitation
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cycle Ergometry + Standard PT/OT (Experimental): The study intervention will include the same standard PT/OT procedures as the control arm (Standard PT/OT alone) with the addition of the Motomed Letto 2 lower extremity cycle ergometry sessions.
  Interventions: Device: Cycle ergometry
- Standard PT/OT alone (No Intervention): The control arm will involve standard PT/OT procedures that patients in the transplant intensive care unit receive routinely, with frequency to be determined by a physical and/or occupational therapist, and may include but are not limited to the following:
  Passive and active upper and lower extremity strength exercises, while in bed, sitting upright, and standing; stretching various muscle groups while supine in bed, sitting upright, and standing; in-bed mobility training including rolling and boosting; transfer training with and without an assistive device; gait training with and without an assistive device; balance exercises while sitting and standing; activities of daily living while sitting and standing; cognitive retraining

INTERVENTIONS:
Device: Cycle ergometry — Lower extremity cycle ergometry, passive and/or active, up to 20 minutes per session, up to 5 sessions per week
  Arms: Cycle Ergometry + Standard PT/OT

SUMMARY:
Critically-ill patients with liver disease are at high risk of developing sarcopenia and intensive care unit (ICU)-acquired weakness, which are associated with mortality and other poor outcomes. Early physical rehabilitation has shown benefit in ICU settings, but has not been studied in ICU patients with acute and chronic liver failure. Cycle ergometry, or stationary cycling in passive and active modes, may be especially beneficial to such patients due to their high prevalence of severe physical deconditioning and variable mentation. The aim of this study is to examine the feasibility, safety, and benefit of cycle ergometry over standard physical and occupational therapy (PT/OT) in critically-ill patients who have acute or chronic liver disease.

DETAILED DESCRIPTION:
A single-blinded randomized controlled trial will be conducted in a transplant intensive care unit (TICU). Eligible adult patients will be enrolled within 72 hrs after TICU admission and randomly allocated to either (1) standard PT/OT care, or (2) PT/OT care and cycle ergometry sessions with trained PT/OT therapists or technicians. The outcome measures, tests of strength and function, will be assessed at baseline, every 14 days, and upon TICU discharge by a blinded PT/OT therapist.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 ≥ years with acute or chronic liver disease admitted to Transplant Intensive Care Unit (TICU), or admitted to TICU following a liver or liver-kidney transplant
* Expected to remain in ICU for ≥ 5 days
* Spoken English fluency

Exclusion Criteria:

* Known primary systemic neuromuscular disease or intracranial process causing increased intracranial pressure
* Lower extremity amputation
* Anticipated death or palliative withdrawal of life support within 5 days
* Cycle ergometer weight limit (135 kg or 297.6 lbs per manufacturer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Functional Status Score for the Intensive Care Unit (FSS-ICU) | Through study completion, average of 1 year
  Standardized assessment tool for functional status in ICU patients. Score ranges from 0 (unable to perform) to 35 (highest function).

SECONDARY OUTCOMES:
Number of participants who experience an adverse event during therapy | Through study completion, average of 1 year
  Total number of participants who experience an adverse event during PT/OT and cycling sessions during course of study
Duration of mechanical ventilation | Through study completion, average of 1 year
  Average number of days on mechanical ventilation
ICU length of stay | Through study completion, average of 1 year
  Average length of stay in days
Number of participants who experience ICU readmission | Through study completion, average of 1 year
  Total number of participants readmitted to ICU during study period

CONTACTS AND LOCATIONS:
Overall Officials: Priyal Patel, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States